CLINICAL TRIAL: NCT04287777
Title: Ph-III Randomized, Multicentric, Controlled , Non-inferiority Trial to Evaluate the Safety and Efficacy of Mupirocin Gel 20 mg/g Versus Mupirocin Ointment 20 mg/g and Placebo in the Treatment of Impetigo in Paediatric Population
Brief Title: Safety and Efficacy of Mupirocin Gel in Children With Impetigo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reig Jofre Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RJ-NBC01
Record Dates: First submitted 2015-10-29; First posted 2020-02-27 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Impetigo
Keywords: Impetigo; Mupirocin; Mupirocin gel; Mupirocin ointment; Impetigo in children
MeSH Terms: conditions — Impetigo | interventions — Mupirocin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mupirocin gel (Experimental): Topical administration of Mupirocin gel 20 mg/g BID for 7 days
  Interventions: Drug: Mupirocin gel
- Mupirocin ointment (Active Comparator): Topical administration of Mupirocin ointment 20mg/g TID for 7 days.
  Interventions: Drug: Mupirocin ointment
- Placebo (Placebo Comparator): Topical administration of Placebo (ointment) TID for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mupirocin gel — Topical administration of Mupirocin gel 20 mg/g BID for 7 days
  Arms: Mupirocin gel
Drug: Mupirocin ointment — Topical treatment of Mupirocin ointment 20 mg/g TID for 7 days
  Other Names: Bactroban
  Arms: Mupirocin ointment
Drug: Placebo — Topical administration of Placebo (ointment) TID during 7 days
  Arms: Placebo

SUMMARY:
The purpose of the study is to show non inferiority in terms of safety and efficacy of topical administration BID (Twice daily) of Mupirocin Gel 20 mg/g compared to topical administration of Mupirocin Ointment 20 mg/g TID (three times daily) (Bactroban) in the treatment of impetigo in paediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 months and 15 years at the signature of informed consent
* Impetigo susceptible to be treated with topical mupirocin and non requiring systemic antibiotic treatment (maximum of 4 different affected areas and no fever).
* Global score of Skin Infection Rating Scale (SIRS) ≥ 4, with positive value (≥ 1) in at least 3 of the 5 categories evaluated.
* Signature of informed consent by parent or legal tutor and, in case of mature minor (12 years or more), signature of informed assent.
* Patient or parent's ability to understand and fulfill with protocol requirements.
* In potentially pregnant patients, negative pregnancy urine test at baseline and use of reliable contraception double barrier methods during the trial.

Exclusion Criteria:

* Allergy to any compound of the trial treatments
* Have received systemic treatment with antibiotics or steroids, during the week prior to the baseline visit.
* Have received topical treatment with corticosteroids, antibiotics or antifungals, during the 48 hours prior to the baseline visit.
* Primary or secondary immunodeficiency.
* Have received cytostatic or immunosuppressive treatment three months prior to baseline.
* Any skin disorder that could interfere with the evaluation of the results of impetigo, such as presence of staphylococcal or streptococcal ecthyma, cellulitis, furunculosis, acute dermatitis, contact dermatitis or impetiginized eczema.
* Diabetes mellitus.
* Infection that, in the investigator's opinion, should be treated with systemic antibiotic.
* Any medical condition which, in the investigator's opinion, contraindicates the subject's participation in the trial.
* Forecast of little cooperation, non-compliance with medical treatment or low credibility.
* Have participated in any clinical investigation with medicine within 30 days prior to basal visit.

Ages: 18 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 467 (Actual)
Dates: Start 2014-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Clinical cure at the end of treatment by SIRS assessed by blind observer | Day 8
  Proportion of subjects with clinical cure at the Day 8 visit, assessed by blind observer, according to criteria described in the Protocol (SIRS < or = 2).
Clinical cure as assessed by the proportion of subjects with no additional antibiotic therapy required to treat impetigo at day 8 | Day 8
  proportion of subjects with no additional antibiotic therapy required to treat impetigo

SECONDARY OUTCOMES:
Clinical cure at the end of follow up by SIRS assessed by blind observer | Day14
  Proportion of subjects with clinical cure at the Day 14 visit, assessed by blind observer, according to criteria described in the protocol (SIRS < or = 2).
Clinical cure as assessed by the proportion of subjects with no additional antibiotic therapy required to treat impetigo at day 14 | Day14
  proportion of subjects with no additional antibiotic therapy required to treat impetigo
Total SIRS score at the end of treatment and follow-up by blind observer | Day 8 and 14
Bacteriology cure at follow-up | Day 14
  Bacteriology eradication at the end of follow-up period according to culture at screening and follow up visits
Clinical cure at the end of treatment and follow-up by investigator | Day 8 and 14
  Proportion of subjects with clinical cure at the Day 8 and Day 14 visits, assessed by investigator, according to protocol criteria.
SIRS total score at the end of treatment and follow-up by investigator | Day 8 and 14
  SIRS total Score at Day 8 and Day 14 visits, assessed by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Raúl De Lucas, Dr., Study Director — Hospital La Paz
Locations (20):
- Spain (20):
  - CAP Torreblanca, Seville, Andalusia
  - CAP La Algaba, Seville, Andalusia
  - CAP Vallcarca-St. Gervasi, Barcelona, Catalonia
  - CAP Corbera de Llobregat, Corbera de Llobregat, Catalonia
  - CAP Amadeu Torner, L'Hospitalet de Llobregat, Catalonia
  - CAP Mossèn Cinto Verdager, L'Hospitalet de Llobregat, Catalonia
  - CAP Florida Nord, L'Hospitalet de Llobregat, Catalonia
  - CAP Rambla Ferran, Lleida, Catalonia
  - CAP Maria Bernades, Viladecans, Catalonia
  - H.U. Sureste, Arganda, Madrid
  - H.U. Fuenlabrada, Fuenlabrada, Madrid
  - CAP Castilla la Nueva, Fuenlabrada, Madrid
  - CAP Pinto, Pinto, Madrid
  - CAP Pozuelo de Alarcón, Pozuelo de Alarcón, Madrid
  - H.U. Infanta Sofía, San Sebastián de los Reyes, Madrid
  - CAP Cea Bermúdez, Madrid
  - Hospital Gregorio MArañón, Madrid
  - CAP Campo de la Paloma, Madrid
  - CAP Aravaca, Madrid
  - CAP La Calesas, Madrid